CLINICAL TRIAL: NCT04862117
Title: Long Term Extension Study of the Safety and Efficacy of Neurostimulation Using a Vagus Nerve Stimulation Device in Patients With Rheumatoid Arthritis
Brief Title: Long Term Extension of Safety and Efficacy of Vagus Nerve Stimulator in Patients With Rheumatoid Arthritis (RA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPM-011
Record Dates: First submitted 2021-02-22; First posted 2021-04-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active stimulation QD (Active Comparator)
  Interventions: Device: SetPoint Medical Neurostimulation of the Cholinergic Anti-inflammatory Pathway System
- Active stimulation QID (Active Comparator)
  Interventions: Device: SetPoint Medical Neurostimulation of the Cholinergic Anti-inflammatory Pathway System

INTERVENTIONS:
Device: SetPoint Medical Neurostimulation of the Cholinergic Anti-inflammatory Pathway System — Active Implantable Vagus Nerve Stimulation device.
  Other Names: SetPoint System

SUMMARY:
Long-term extension of a multi-site, first-in-human study to assess safety and efficacy of an active implantable Vagus Nerve Stimulation (VNS) device in adult patients with active moderate-to-severe rheumatoid arthritis who have had an incomplete response or intolerability to at least two biologic and/or targeted synthetic DMARDs having at least two different mechanisms of action

DETAILED DESCRIPTION:
A multicenter, extension study to assess long term safety and efficacy of an active implantable VNS device in adult patients with rheumatoid arthritis. The study is uncontrolled and randomized, where the sites and subjects are blinded to treatment until completion of the parent study. Subjects who were randomized to the inactive device group in the parent study are re-randomized to receive active vagus nerve stimulation either 1 min QD or 1 min QID. Subject who were randomized to the active device groups remain on their assigned treatment (1 min QD, 1 min QID).

Study treatment in SPM-011 begins at the Day 0 Visit. At the Day 0, Week 1, 2, 3, 4 and 5 Visits, all subjects are given the opportunity to have the output current of their implant adjusted to the maximum level tolerated.

From Week 5 onward, subjects will receive their maximally tolerated output current as 1 min QD or 1 min QID treatment.

Follow up assessment visits occur at Week 8, Week 12, Months 6, 9, 12, 18, 24, 30, 33 and 36. Subjects are assessed for safety and durability of response throughout the follow up period. If the subject's symptoms or RA disease worsens, additional concomitant medications are allowed for treatment of their RA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have enrolled and completed 12 weeks of treatment in Study SPM-008
2. Women of childbearing potential must not be pregnant and must agree to use a reliable method of contraception throughout the study

Exclusion Criteria:

1. Inability to provide consent
2. An adverse event during Study SPM-008 which precludes participation in this study
3. Any condition per the investigator's clinical judgement that precludes participation in the study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2026-12-08 (Estimated); Study Completion 2026-12-08 (Estimated)

PRIMARY OUTCOMES:
Incidence rates of Adverse Events | Enrollment through Month 36 (End of Study)
  Treatment-emergent incidence rates of Adverse Events, Adverse Device Effects, Serious Adverse Events, Serious Adverse Device Effects, Unanticipated Adverse Device Effects, and Unanticipated Serious Adverse Device Effects

SECONDARY OUTCOMES:
Change in Disease Activity Score (DAS) 28 - C-reactive protein (CRP) | Day 0 through Month 12
  Mean change in Disease Activity Score (DAS) 28 - C-reactive protein (CRP)
American College of Rheumatology (ACR) 20, 50 and 70 response rates | Day 0 through Month 12
  Percentage of subjects meeting American College of Rheumatology (ACR) 20, 50 and 70 response status
European League Against Rheumatism (EULAR) response rates | Day 0 through Month 12
  Percentage of subjects meeting European League Against Rheumatism (EULAR) response status of Good, Moderate and None
Disease Activity Score (DAS) 28 - C-reactive protein (CRP) remission rate | Day 0 through Month 12
  Percentage of subjects meeting Disease Activity Score (DAS) 28 - C-reactive protein (CRP) remission

CONTACTS AND LOCATIONS:
Overall Officials: Alan Kivitz, MD, Principal Investigator — Altoona Center for Clinical Research
Locations (4):
- United States (4):
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Northwell Health, Great Neck, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania